CLINICAL TRIAL: NCT04751864
Title: Fisher Wallace Brain Stimulation & Generalized Anxiety Study
Brief Title: Brain Stimulation & Generalized Anxiety Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: ProofPilot (Industry)
Collaborators: Fisher Wallace (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2503
Record Dates: First submitted 2020-11-09; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Anxiety; Generalized Anxiety Disorder; Generalized Anxiety
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Participants randomized into Sham and Active device arms for four weeks. At the week 5 crossover, participants in sham arm receive active device.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Arm (Experimental): Participants receive active device for the full 8 week study
  Interventions: Device: Cranial Electrotherapy Stimulator (CES) Device
- Sham Arm (Sham Comparator): Participants receive sham device for the first 4 weeks, and then at the week 5 cross over, receive the active device.
  Interventions: Device: Cranial Electrotherapy Stimulator (CES) Device

INTERVENTIONS:
Device: Cranial Electrotherapy Stimulator (CES) Device — Fisher Wallace Cranial Electrotherapy Stimulator (CES) Device

SUMMARY:
Examine the safety and effectiveness of the Fisher Wallace Cranial Electrotherapy Stimulator (CES) Device on Generalized Anxiety Disorder using two (2) 20-minute per day treatment sessions over eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 21
* US resident
* Can receive packages to their home via UPS/Fedex/USPS
* Licensed Physician Diagnosis of Generalized Anxiety Disorder
* Beck Anxiety Inventory Score between 8 and 25
* Read/write English
* Have not contemplated suicide in the past year
* Not been institutionalized for mental health issues.
* Not currently experiencing problems with alcohol or drug abuse
* Can commit to not drinking alcohol 4 hours before bedtime for the duration of the study
* Can commit to two (2) 20 minute sessions per day for 8 weeks
* Not under medical supervision for serious medical condition
* Not currently being treated for or suspect a mental health issue
* Has not used a brain stimulation treatment in one year
* No suspected or known history of heart disease
* No pacemaker, or any form of medical electronics, including but not limited to a deep - brain stimulator, electronic stent, etc.
* Not taking opioids
* Are a resident of states in which we have licensed medical professionals
* Does not have any co-occurring significant psychiatric disorder that would impair - participant's particationion.
* Does not use any illicit drugs
* Not participating in any other anxiety study
* Not taking medications affecting the nervous system (e.g. psychiatric medications)
* Not taking hypnotics or any sleep aid or marijuana (in any form)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-06-21 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Anxiety Inventory (BAI) Score | baseline versus week 4
  The Beck is a 21 item self-reported scale measuring anxiety

SECONDARY OUTCOMES:
Change in Promise Sleep-SD | baseline versus week 4
  Change in self reported sleep quality
Change in Patient Health Questionnaire - 8 (PHQ-8) | baseline versus week 4
  self reported depression symptoms
Change in Beck Anxiety Inventory (BAI) Score | week 4 versus week 8
  The Beck is a 21 item self-reported scale measuring anxiety
Device safety, tolerability and adherence as measured by SAFTEE | baseline versus week 8
  The SAFTEE is a self reported measure of side effects associated with mental health treatments

CONTACTS AND LOCATIONS:
Locations (1):
- ProofPilot (Remote Virtual Trial), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No